CLINICAL TRIAL: NCT05819489
Title: A Comparison of Dynamic Vision & Balance Between College Athletes & Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: California State University, Northridge (Other)
Responsible Party: Principal Investigator, Aimie Kachingwe, Primary Investigator, California State University, Northridge
Other Study IDs: IRB-FY23-271
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Head Injury; Sport Injury; Concussion, Brain
MeSH Terms: conditions — Craniocerebral Trauma; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dynamic Vision Testing — Dynamic Vision Testing (Bertec Vision Advantage System) and Balance Error Scoring System Assessment tool and computerized tests designed to evaluate postural stability and vestibulo-ocular reflex (VOR) function while assisting with return to play decision after a sports-related concussion.
  Other Names: Balance Error Scoring System Assessment

SUMMARY:
The purpose of this study is to determine the value of including dynamic vision testing into California State University, Northridge (CSUN) Athletics' established concussion protocol. The study's hypotheses are 1) dynamic vision testing will reveal vision impairments right after a person sustains a concussion, 2) these impairments may still be present upon clearance to return to play.

DETAILED DESCRIPTION:
The subjects of interest are CSUN student-athletes who give consent to participate in the study. Dynamic vision will be assessed through the administration of the Dynamic Visual Acuity (DVA) test and the Gaze Stabilization Test (GST). Additionally, the 6-condition Balance Error Scoring System (BESS), which is currently a component of CSUN's established concussion protocol, will be administered to assess balance impairments. This cluster of tests will be administered three times per athlete: (1) during preseason to establish baseline measures, (2) acutely post-concussion once the athlete subject has been cleared by the team physician for return to exercise, and (3) when cleared to return to sport. The results will be used to evaluate whether or not dynamic vision results have returned to baseline by the time that CSUN Athletics clears the athlete to "Return to Play."

ELIGIBILITY:
Inclusion Criteria:

* California State University Northridge athletes
* Participants are able to give consent to participate in the study
* Completion of preseason testing for the 6-condition, BESS, DVA, GST with the research team
* Sustained a concussion as diagnosed by the medical staff during the 2020-2021 season of play.
* Sampling of convenience on a volunteer basis

Exclusion Criteria:

* Athletes with preseason baseline tests on BESS or DVA that are not within the normative value range for an unimpaired individual.
* The initial 6- condition BESS score is >20 errors
* The subject is unable to attain a minimum of 85 degrees per second of horizontal head rotation when performing the DVA test.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Due to COVID-19 and the uncertainty of which teams will be competing during the academic year, our subject pool will potentially come from any athlete who provides consent from an equal number of men's and women's teams who are competing that semester.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
6 Condition BESS | August 15, 2021 - August 15, 2024
  Number of errors and time subject was able to hold position Number of errors and time subject was able to hold position Number of errors and time subject was able to hold position

SECONDARY OUTCOMES:
Gaze Stabilization Test (GST) | August 15, 2021 - August 15, 2024
  Maximum head velocity in degrees/second

OTHER OUTCOMES:
Dynamic Visual Acuity (DVA) | August 15, 2021 - August 15, 2024
  Log of minimal angle resolvable units (LogMAR). The number of lines on an eye chart that are lost with head moving.
  (DVA) compared to the head steady condition, known as static visual acuity (SVA)

CONTACTS AND LOCATIONS:
Overall Officials: Aimie Kachingwe, Dr., Principal Investigator — CSUN; Margaret Roller, Dr., Principal Investigator — CSUN
Locations (1):
- California State University, Northridge, Jacaranda Hall 1578, 1576, 1574, Northridge, California, United States

IPD SHARING:
Plan to Share IPD: No